CLINICAL TRIAL: NCT06907901
Title: Reliability Analysis of the Postural Habits and Awareness Scale (PHAS) in Patients With Postural Hyperkyphosis
Brief Title: Reliability of PHAS in Postural Hyperkyphosis
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Assoc. Prof., Istanbul University - Cerrahpasa
Other Study IDs: aza_isu1
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-03

CONDITIONS: Postural Kyphosis; Spine; Assessment, Self
Keywords: Hyperkyphosis; Postural Habits; Postural Awareness; Psychometric Analysis; Spinal Deformity; Postural Evaluation
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyperkyphosis Group: Participants diagnosed with postural hyperkyphosis completing the PHAS and KSSA for reliability analysis.
  Interventions: Behavioral: PHAS Assessment

INTERVENTIONS:
Behavioral: PHAS Assessment — Participants will complete the Postural Habits and Awareness Scale (PHAS) to assess postural awareness and habits. The scale will be administered twice, two weeks apart, to evaluate reliability.

SUMMARY:
This observational, cross-sectional study aims to evaluate the reliability of the Postural Habits and Awareness Scale (PHAS) in patients with postural hyperkyphosis. The PHAS is designed to assess individuals' postural awareness and habits through four subscales. A total of 128 participants diagnosed with postural hyperkyphosis will complete the PHAS and the Kyphosis-Specific Spinal Appearance Questionnaire (KSSA). Test-retest reliability will be assessed by reapplying the PHAS after two weeks. Internal consistency, test-retest reliability, and concurrent validity will be analyzed. The study aims to provide a valid and reliable tool for evaluating postural awareness in clinical practice and future rehabilitation studies.

DETAILED DESCRIPTION:
This study is designed to assess the reliability of the Postural Habits and Awareness Scale (PHAS) in individuals diagnosed with postural hyperkyphosis. Postural hyperkyphosis is increasingly common due to sedentary lifestyles, prolonged sitting, and technological device use, leading to significant postural deviations and musculoskeletal complaints. Early detection and management of postural habits are essential to prevent long-term spinal deformities and functional limitations.

The PHAS was developed to systematically evaluate individuals' postural awareness and habits in daily life, focusing on factors that contribute to poor posture and spinal alignment. The scale assesses dimensions such as postural habits, awareness of posture-disturbing factors, positional awareness, and ergonomic considerations. However, its psychometric properties, particularly reliability in hyperkyphotic patients, have not yet been established.

This observational, cross-sectional methodological study will employ standardized psychometric methods to analyze the internal consistency and test-retest reliability of the PHAS. The scale's ability to produce stable and consistent results over time will be tested through repeated administration. Additionally, concurrent validity will be examined by comparing PHAS scores with the Kyphosis-Specific Spinal Appearance Questionnaire (KSSA), which measures patients' perception of their spinal deformity.

The findings will provide valuable insights into the scale's utility for clinical and research purposes. Establishing PHAS as a reliable tool could allow physiotherapists, ergonomists, and healthcare professionals to objectively assess postural habits and awareness, design personalized rehabilitation programs, and monitor treatment outcomes. Furthermore, the scale could be integrated into preventive strategies aimed at improving postural control and spinal health in both clinical practice and community settings.

Research Team:

Assoc. Prof. Dr. Ayşe Zengin Alpözgen (Principal Investigator) PhD. PT Kübra Kardeş (Istinye University) MSc PT Selin Uz Tunçay (Istanbul University-Cerrahpasa) MSc PT Merve Koyuncu Cenikli (Istanbul University-Cerrahpasa)

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 65 years
* Diagnosed with postural hyperkyphosis (Cobb angle ≥ 50° confirmed by clinical and radiological evaluation)
* Ability to perform daily activities independently
* Voluntary participation and signed informed consent

Exclusion Criteria:

* Presence of scoliosis or other spinal deformities
* Kyphosis due to severe osteoporosis or pathological fractures
* Diagnosis of ankylosing spondylitis or other inflammatory spinal diseases
* Functional limitations due to acute or chronic pain
* Previous postural awareness training or spinal rehabilitation within the last 6 months
* Cognitive impairment or severe psychiatric disorder preventing independent questionnaire completion

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals diagnosed with postural hyperkyphosis. Participants will include patients aged 8 to 65 years who have been clinically and radiologically confirmed to have postural hyperkyphosis with a Cobb angle of 50° or higher. All participants are expected to be capable of performing daily activities independently.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Reliability of the Postural Habits and Awareness Scale (PHAS) | 2 weeks
  Internal consistency will be evaluated using Cronbach's Alpha. Test-retest reliability will be assessed by calculating the Intraclass Correlation Coefficient (ICC) between two PHAS administrations. The PHAS consists of 19 items, each scored on a 5-point Likert scale (total score range: 19 to 95). Higher scores indicate better postural habits and awareness. Higher ICC values indicate better reliability.

SECONDARY OUTCOMES:
Kyphosis-Specific Spinal Appearance Questionnaire (KSSAQ) | Baseline
  The KSSAQ is a 10-item, 5-point Likert scale (range: 1 to 5 per item, total score range: 10 to 50) designed to assess patients' perception of their spinal appearance related to thoracic hyperkyphosis. Higher scores indicate worse perceived deformity and greater concern about appearance. The correlation between PHAS and KSSAQ scores will be calculated to determine concurrent validity.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Zengin Alpözgen, Assoc. Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided